CLINICAL TRIAL: NCT02674776
Title: A Clinical Trial About the Efficacy and Safety of HuZhen Capsule in Treating Patients With Acute Gout: A 72 Hours, Multi-center, Randomized, Double-blind, Parallel Placebo Compared Clinical Trial
Brief Title: Efficacy and Safety of HuZhen Capsule for Treatment of Patients With Acute Gout
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Quan Jiang (Other)
Responsible Party: Sponsor-Investigator, Quan Jiang, Director and Professor of Rheumatology Devision, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013003P3A03
Record Dates: First submitted 2016-01-28; First posted 2016-02-04 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Acute Gout

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HuZhen Capsule (Experimental): The main elements of HuZhen Capsule include Polygonum cuspidatum, Ligustrum lucidum etc.
  Interventions: Drug: HuZhen Capsule
- Placebo Capsule (Placebo Comparator): Placebo appearance, content color and taste should be consistent with HuZhen Capsule.
  Interventions: Drug: Placebo Capsule

INTERVENTIONS:
Drug: HuZhen Capsule — Patients should take 4 tablet once and 3 times per day for 3 days.
  Other Names: capsule A
  Arms: HuZhen Capsule
Drug: Placebo Capsule — Patients should take 4 tablet once and 3 times per day for 3 days.
  Other Names: capsule B
  Arms: Placebo Capsule

SUMMARY:
This study is a multi-center, double-blind, randomized, parallel controlled trial. Patients with acute gout will be enrolled and randomly allocated into 2 groups: HuZhen capsule treatment group and Placebo control group. Randomization codes were established by the biostatistician. Observe will be followed for 3 days (72 hours) after the onset. Change of VAS score from baseline, proportion of improvement with damp-heat retention, change in C-reactive protein (CRP) and erythrocyte sedimentation rate ( ESR) from baseline, change in white blood cell count in whole blood cell analysis from baseline, and the number of adverse events will be monitored and compared between each groups.

DETAILED DESCRIPTION:
The test group will be given HuZhen capsule 1.6g three times per day,the control group will be given placebo 1.6g three times per day. The invention will last 3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Score is equal to or larger than 40cm on the 0-100cm VAS pain scale.
2. Acute attack of gout no longer than 2 days.
3. Participant with acute gout is diagnosed as "damp-heat retention" by Traditional Chinese medicine.
4. Age 18-65 years with informed consent.

Exclusion Criteria:

1. Chronic gouty arthritis.
2. Pseudogout, acute rheumatic fever and suppurative arthritis, traumatic arthritis, erysipelas, meander rheumatism and other arthritis.
3. Anti-inflammatory medication for the treatment of acute gout.
4. Pregnant or breastfeeding women.
5. History of severe allergy, including diclofenac sodium.
6. Serum creatinine is higher than the upper normal limit. ALT or AST is higher than the upper normal limit for two times.
7. Fever ( T>38.5 ℃)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change of VAS (visual analog scale) score from baseline to 72 Hours after onset | baseline,72 hours

SECONDARY OUTCOMES:
Proportion of participants with improvement in acute gout at 72 hours post-dose using the criteria for the diagnosis of damp-heat retention | 72 hours
  Refer to the"Guidline for Clinical Study of New Chinese Medicines "
Change in C-reactive protein (CRP) from baseline to 72 hours | baseline,72 hours
  Units of Measure:mg/L
Change in erythrocyte sedimentation rate ( ESR) from baseline to 72 hours | baseline,72 hours
  Units of Measure:mm/hour
Change in white blood cell count in whole blood cell analysis from baseline to 72 hours | baseline,72 hours
The number of adverse events related to treatment | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Quan, Doctor, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided